CLINICAL TRIAL: NCT04226014
Title: Score of Echogenicity and Pancreatic Echo-endoscopy
Brief Title: Observational Cohort of Pancreatic Echo-endoscopy
Acronym: OBELIX
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Saint Joseph Saint Luc de Lyon (Other)
Collaborators: Clinique du Val d'ouest (Unknown)
Responsible Party: Sponsor
Other Study IDs: OBELIX
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Metabolic Syndrome; Obesity; Hepatic Steatosis
Keywords: pancreatic echogenecity; Hepatic Steatosis; Metabolic Syndrome; Obesity
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Fatty Liver | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with echo-endoscopic ultrasound of the pancreas: Patients requiring endoscopic ultrasound of the pancreas were included in the cohort.
  Interventions: Procedure: Endoscopic ultrasound

INTERVENTIONS:
Procedure: Endoscopic ultrasound — Echo-endoscopy ultrasound is an examination that presents little risk. However, any medical act, exploration, intervention even conducted under conditions of competence and safety in accordance with current data of medicine and the regulations in force, conceals a risk of complications. In particular, esophageal perforations can occur. They are often favored by underlying lesions (tumor, diverticulum, anatomical variants ...). Other complications are possible such as cardiovascular, respiratory or infectious disorders, as with any anesthesia.

SUMMARY:
Metabolic syndrome is defined by the presence of at least two of the following five criteria: abdominal perimeter> 94 cm in men, 80 cm in women, high triglycerides, low HDL cholesterol, HTA and hyperglycemia.

The metabolic syndrome can lead to ultrasound hepatic steatosis in 20 to 40% of cases depending on the population studied (overweight vs obesity). What is the impact of this syndrome on pancreatic echogenicity?

DETAILED DESCRIPTION:
Little is known about the pathogenesis of the fatty pancreas. Fat can replace acinar cells and / or pancreatic endocrine cells (1). To date, there are no biomarkers allowing the detection of a fatty pancreas. It appears that older age, male, obesity, alcohol consumption, high triglycerides, high ALT, diabetes or insulin resistance, fatty liver and metabolic syndrome are risk factors for a fatty pancreas (2,3,4).To the investigator's knowledge, these different factors have not been evaluated on the impact of pancreatic echogenecity in endosonography. The objective of this study is to correlate the factors making up the metabolic syndrome with pancreatic echogenecity.

ELIGIBILITY:
Inclusion Criteria:

* any consecutive patient, having a high echo-endoscopy
* for an extra pancreatic cause, such as the search for a cholelithiasis, (the pancreas will be studied completely)
* for esophageal pathologies, (the pancreas will be studied completely)
* for gastric pathologies, (the pancreas will be studied completely)
* for cystic lesions of the pancreas (pancreas studied upstream and downstream)
* for submucosal tumors (esophageal / gastric / duodenal)
* for abdominal pain of undetermined origin

Exclusion Criteria:

* Patients with pancreatic and / or tissue damage with dilated wirsung canal and / or acute or chronic pancreatitis.
* Patients having contraindication to general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient receiving a high echo-endography meeting the inclusion criteria will be included.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Correlation of the pancreatic echogenicity by endoscopic ultrasound with the metabolic syndrome | During the reading of the echo-endoscopic procedure
  Three categories of echogenicity have been defined. The presence of one or more factors of the metabolic syndrome was correlated with the category of pancreatic echogenicity defined by the experts

SECONDARY OUTCOMES:
Comparaison of the echogenicity of the pancreas with respect to the liver and to the spleen will be made. | During the reading of the echo-endoscopic procedure
  The pancreatic echogenicity score will be assessed with the following criteria
  1. The visibility of Wirsung in three categories: excellent, average, poor
  2. that of the contours in 3 categories good or average or poor visualization of the splenic vein
  3. that of the parenchyma in 3 categories: normal, brilliant, not too obstructing the visualization of the Wirsung and the splenic vein, very promising embarrassing the visualization of the Wirsung and the splenic vein
  4. with in addition a -heterogeneous or - homogeneous item for the parenchyma.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie MARION-AUDIBERT, MD, PhD, Principal Investigator — Clinique du Val d'ouest
Locations (5):
- France (5):
  - Polyclinique du Beaujolais, Arnas
  - Clinique du Val d'Ouest, Écully
  - Hôpital privé Jean Mermoz, Lyon
  - Clinique du Trocadéro, Paris
  - Clinique des Portes du Sud, Vénissieux